CLINICAL TRIAL: NCT05922098
Title: To Explore the Effect of Improved Modified Care Meals to Improving the Quality Of Life of the Pre-Frailty Chewing Disorders of the Older Adult
Brief Title: Improved Modified Care Meals to Improving the Quality Of Life of the Pre-Frailty Chewing Disorders of the Older Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, WangJiaJie, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: WangJiaJie
Record Dates: First submitted 2023-05-02; First posted 2023-06-28 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Food Selection; Quality of Life; Chewing Disease; Satisfaction
MeSH Terms: conditions — Food Preferences; nigropallidal encephalomalacia; Personal Satisfaction | interventions — Aging

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Texture Modified Foods Manual for chewing dysfunctions (including IDDSI)
  Interventions: Other: Texture Modified Foods Manual for chewing dysfunctions in older adult
- control group (No Intervention): Traditional Soft Food Care Manual

INTERVENTIONS:
Other: Texture Modified Foods Manual for chewing dysfunctions in older adult — Texture Modified Foods Manual for chewing dysfunctions (including IDDSI)
  Arms: experimental group

SUMMARY:
In 2020, we have entered an aging society. During the aging process, the body will decline with age, and the muscles will decrease, which will affect the swallowing muscles, causing chewing and swallowing difficulties are very common. Difficulty masticating is associated with problems with real teeth, dentures, and oral health disease, and is associated with infection, pain, inadequate nutritional intake, affected appearance, decreased quality of life, and mortality.

At present, Taiwan mostly provides the elderly with shredded food, cooked soft and rotten food, or whipped food. However, when the food is mashed or shredded, the original color, fragrance, and taste of the food will be lost. It cannot change the appetite of the elderly, and it will reduce the satisfaction of the elderly's meal, and there will still be risks of insufficient food intake and uneven nutrition. Appearance or taste can improve the satisfaction and quality of life of the elderly, improve the health needs of nutrition, and allow a variety of choices when eating to change the current situation of traditional whipped food and shredded meals.It is expected that the quality of life, nutritional status, and meal satisfaction of the pre-frail elders with masticatory difficulties will be significantly higher than those of the control group if the subjects receive care meals, which can be used as a reference for the daily care of the elderly with masticatory disorders in the future.

ELIGIBILITY:
Inclusion Criteria:

* Elderly over 65 years old.
* Elders who are pre-frail cases after the five assessments of frailty and who are abnormal after the chewing test.
* Clear awareness, willing to accept visitors, able to communicate in Chinese and Taiwanese.
* Ability to express food appearance and taste.
* Those who eat by mouth.

Exclusion Criteria:

* Elderly with dementia (certified by medical records and disability handbook).
* Elderly people who have swallowing disorders in the throat stage after being screened by the modified water swallowing test.
* Visually impaired and no primary caregiver to assist the program implementer.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Geriatric oral health assessment index，GOHAI | 10-20mins
  Total score is 64 points, with higher scores indicating poorer oral health
Oral Health Assessment Tool ，OHAT | 10-20mins
  Total score is 16 points, with higher scores indicating poorer oral health
Oral health impact profile，OHIP | 10-20mins
  Total score is 56 points, with higher scores indicating poorer oral health
Meal satisfaction seven-item questionnaire | 5-10mins
  full score 35, minimum score 5 points.

SECONDARY OUTCOMES:
Mini Nutritional Assessment - MNA Elderly, | 5-10mins
  Less than or equal to 7 points for malnutrition; 8-11 points for high-risk groups of malnutrition; 12 points for normal.

CONTACTS AND LOCATIONS:
Overall Officials: Wang JiaJie, Principal Investigator
Locations (1):
- WangJiaJie, Hualien City, Taiwan